CLINICAL TRIAL: NCT02491957
Title: Impact of LOFT Therapy™ on Breast Cancer Survivors: A Pilot Study
Brief Title: Impact of LOFT Therapy™ on Breast Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kathy Miller (Other)
Responsible Party: Sponsor-Investigator, Kathy Miller, Professor of Medicine and Sheila D. Ward Scholar, Indiana University School of Medicine
Organization: Indiana University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IUSCC-0539
Record Dates: First submitted 2015-06-02; First posted 2015-07-08 (Estimated); Last update posted 2018-08-13 (Actual); Status verified 2018-08

CONDITIONS: Breast Neoplasms
Keywords: Energy Expenditure; Physical Endurance; Muscle Stength; Metabolism
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- LOFT Therapy (Experimental): LOFT therapy twice weekly for 4 weeks
  Interventions: Other: LOFT Therapy

INTERVENTIONS:
Other: LOFT Therapy — LOFT Therapy™ will be performed 2 times a week for 4 weeks a total of 8 sessions. The patient will be wrapped with fabric cuffs, on up to four limbs. The cuffs are applied to the widest part of the biceps and upper thighs at pressures between 80-100 mmHg with minimal venous encroachment. The patients will ride a recumbent bike for 18 total minutes of sub-maximal exertion (up to 70% repetition maximum ), with the option of up to 2 periods of 15-second higher intensity exertions as tolerated, followed by individualized respiratory recovery periods determined by the relative decrease in breathing effort.
  The 18-minute session will be preceded by a two-minute compression check, where the wraps will be adjusted based on any signs or symptoms of nerve or vessel impingement.

SUMMARY:
The purpose of this study is to evaluate the safety and feasibility of LOFT Therapy in breast cancer survivors. In a previous study, the investigators found that many patients are more debilitated at diagnosis than previously recognized. Both chemotherapy and anti-estrogen therapy have a large effect. Within 6 months patients replace muscle with fat leading to a significant reduction in muscle power and endurance. Our data suggests that common exercise recommendations for at least 150 minutes of exercise a week would be far beyond many of our patients' physical ability after therapy, leading to the soreness, injury, frustration, and early discontinuation (or failure to initiate an exercise program in the first place). The degree of muscle loss seen in our patients is similar to that documented in US astronauts after long-term space flight. Our collaborator Dr. Yvonne Cagle, retired USAF flight surgeon, noted that the cosmonauts were in better shape (had less muscle atrophy) than the astronauts. This difference was more than could be explained by the rigorous Russian exercise program. The only key distinction was the compressive, "penguin suits" used by the Russians. This observation lead Dr. Cagle to develop a technique called low intensity, off loaded-compressive therapy (LOFT) to replicate the impact of the Russian penguin suits for patients who were debilitated, whether by space flight or by chronic conditions such as arthritis, Parkinson's disease, and multiple sclerosis. The LOFT method does not require excessive exertion or strain on the joints. In field observations, LOFT therapy improved muscle strength, muscle mass, endurance, sleep quality, and fatigue. This pilot study is the first to evaluate the safety, feasibility, and biologic impact of LOFT on breast cancer survivors.

DETAILED DESCRIPTION:
Objectives This pilot trial will provide feedback on the feasibility and impact of LOFT in breast cancer survivors. The investigators will also explore the relationship of the LOFT intervention to changes in insulin resistance, growth hormone levels, body mass index, patient reported physical activity, fatigue, and overall quality of life.

Primary Objective Evaluate the safety and feasibility of LOFT training in breast cancer survivors (< 3 years from diagnosis) treated with either chemotherapy and/or anti-estrogen therapy.

Secondary Objectives

1. Estimate the effect size of LOFT training on muscle power, endurance, daily activity, fatigue, and quality of life.
2. Estimate the effect of short-term LOFT training on biochemical parameters of inflammation, metabolism, anabolic hormone secretion, and bone turnover.

LOFT Therapy™ Summary LOFT Therapy™ is a form of exercise that requires less energy for movement. LOFT Therapy™ will be performed 2 times a week for 4 weeks a total of 8 sessions. The patient will be wrapped with fabric cuffs, on up to four limbs. The cuffs are applied to the widest part of the biceps and upper thighs at pressures between 80-100 mmHg with minimal venous encroachment. The patients will ride a recumbent bike for 18 total minutes of sub-maximal exertion (up to 70% repetition maximum ), with the option of up to 2 periods of 15-second higher intensity exertions as tolerated, followed by individualized respiratory recovery periods determined by the relative decrease in breathing effort.

The 18-minute session will be preceded by a two-minute compression check, where the wraps will be adjusted based on any signs or symptoms of nerve or vessel impingement. Patients will undergo an intake and outtake assessment with each session to collect subjective data and patient feedback. Two compression sessions will be conducted for 4 weeks, for a total of 8 sessions.

This study will enroll 15 patients. A 20% dropout rate for this group was taken into consideration so the investigators assume analysis will be done on at least 12 patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with stage 0-III breast cancer within the past 3 years
* Must have completed local therapy for their breast cancer
* Must have received systemic therapy for their breast cancer (anti-estrogen and/or chemotherapy)
* Chemotherapy must be complete prior to entry
* Anti-estrogen therapy may be ongoing
* Ambulatory without assistive devices
* No orthopedic restrictions or neurologic deficits that would limit ability to complete the Power Protocol (based on the opinion of the investigator)
* No requirement for supplemental O2
* No unstable angina, regular use of nitroglycerin for exertional angina, or MI within the last 12 months
* No local or distant recurrence of their breast cancer
* No active lymphedema
* No history of hemorrhagic stroke
* No Heparin or Coumadin Use
* No symptomatic peripheral vascular obstructions
* No active gallbladder disease
* No active kidney stones
* No active gout
* No active diverticulitis
* No pituitary diseases or growth
* Able to provide written informed consent and authorization for release of health information
* Able to commit to LOFT training 2 times/week for 4 weeks

Exclusion Criteria:

* Inability to meet one of the inclusion criteria above.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-07-28 (Actual); Primary Completion 2018-03-29 (Actual); Study Completion 2018-03-29 (Actual)

PRIMARY OUTCOMES:
Feasibility of LOFT therapy in breast cancer survivors (< 3 years from diagnosis) treated with either chemotherapy and/or anti-estrogen therapy | Change from pre-LOFT therapy (baseline) to post-LOFT therapy (5 weeks after baseline)
  Analysis of the modified intent-to-treat population defined as patients with at least 1 post-baseline measurement as well as eligible patients who decline participation, reason for refusal, and number of enrolled patients who do not complete all LOFT training sessions

SECONDARY OUTCOMES:
Safety of LOFT intervention in this population patient reported adverse events | Assessed at each session and throughout the intervention
  Assessed by patient reported adverse events
Heart rate | Change from pre-LOFT therapy (baseline) to post-LOFT therapy (5 weeks after baseline)
Power per body weight (muscle power) | Change from pre-LOFT therapy (baseline) to post-LOFT therapy (5 weeks after baseline)
Endurance | Change from pre-LOFT therapy (baseline) to post-LOFT therapy (5 weeks after baseline)
  Assessed by patient self-report
Daily activity | Change from pre-LOFT therapy (baseline) to post-LOFT therapy (5 weeks after baseline)
  Measured by Physical Activity Report questionnaire
Fatigue | Change from pre-LOFT therapy (baseline) to post-LOFT therapy (5 weeks after baseline)
  Measured by BFI questionnaire
Quality of life | Change from pre-LOFT therapy (baseline) to post-LOFT therapy (5 weeks after baseline)
  Measured by FACT-B questionnaire
Biochemical parameters of chronic inflammation | Change from pre-LOFT therapy (baseline) to post-LOFT therapy (5 weeks after baseline)
  Blood samples
Biochemical parameters of metabolism and insulin homeostasis | Change from pre-LOFT therapy (baseline) to post-LOFT therapy (5 weeks after baseline)
  Blood samples
Anabolic hormone secretion | Change from pre-LOFT therapy (baseline) to post-LOFT therapy (5 weeks after baseline)
  Blood samples
Biochemical parameters of bone turnover | Change from pre-LOFT therapy (baseline) to post-LOFT therapy (5 weeks after baseline)
  Blood samples

CONTACTS AND LOCATIONS:
Overall Officials: Kathy Miller, MD, Principal Investigator — Indiana University School of Medicine
Locations (2):
- United States (2):
  - Indiana University Health Hospital, Indianapolis, Indiana
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana